CLINICAL TRIAL: NCT03398278
Title: An Open-label, Single Dose, Randomised, Cross-over Study to Determine the Fasted State Pharmacokinetics of Oxycodone From Oxycodone Tamper Resistant (OTR) Tablet 40 mg and OXYCONTIN® Tablet 40 mg in Chinese Subjects With Chronic Pain
Brief Title: OTR Tablet 40 mg Fasted-state Bioequivalence Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mundipharma (China) Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ONF16-CN-102
Record Dates: First submitted 2016-07-26; First posted 2018-01-12 (Actual); Results first posted 2019-10-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Receptors, Oxytocin; Tablets; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxycodone Tamper Resistant (Experimental): Oxycodone Tamper Resistant (OTR) Tablet 40 mg
  Interventions: Drug: Oxycodone Tamper Resistant
- OXYCONTIN® (Active Comparator): OXYCONTIN® Tablet 40 mg
  Interventions: Drug: OXYCONTIN®

INTERVENTIONS:
Drug: Oxycodone Tamper Resistant — Orally taking Oxycodone Tamper Resistant 40mg in fast state
  Other Names: Oxycodone Tamper Resistant (OTR) Tablet 40 mg
  Arms: Oxycodone Tamper Resistant
Drug: OXYCONTIN® — Orally taking OXYCONTIN® 40mg in fast state
  Other Names: OXYCONTIN® Tablet 40 mg
  Arms: OXYCONTIN®

SUMMARY:
This is an open-label, single dose, randomised, cross-over study to confirm the bioequivalence (BE) of OTR tablet 40 mg and OXYCONTIN tablet 40 mg in a fasted state in Chinese subjects with chronic pain

DETAILED DESCRIPTION:
In this BE study, subjects with histories of chronic pain are chosen as the target population.

Inclusion/exclusion criteria are strictly defined to reduce the potential variation of the PK data.

Single dose design is chosen per Food and Drug Administration (FDA)/WHO guideline on bioavailability (BA)/BE studies for modified-release products.

As a general rule, cross-over design is applied in the study to decrease the inter-individual variations between the two cohorts. A washout period lasting for at least 7 half-lives of the investigational medicine is needed to eliminate the drug residual from the previous period7. The elimination half-life of oxycodone from OTR is 4.5 hours, and a 6-day washout period is sufficient to achieve the aim.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese male or female subjects with histories of chronic pain regardless of the aetiology, aged 18-55 years both inclusive
2. The average pain over the last 24 hours should be scored < 4 assessed with Numeric Rating Scales (NRS), when not receiving analgesics. The pain condition has been kept stable at least in the past 7 days prior to entering into the screening and is expected to be stable during the study duration
3. Body weight ≥45 kg and a body mass index (BMI) ≥18 and ≤28 kg/m2
4. Karnofsky score of Performance Status ≥70
5. Willing to take all the food supplied while the subject is in the study unit
6. Be able to read, understand, and sign written Informed Consent Form (ICF) prior to study participation and be willing to follow the protocol requirements
7. Willing to use adequate and highly effective methods of contraception throughout the study. A highly effective method of birth control is defined as one which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as sterilisation, implants, injectables, some Intrauterine Device (IUD), sexual abstinence, or vasectomised partner
8. Female subjects, including those up to less than one year post-menopausal, must have a negative serum pregnancy test and be non-lactating

Exclusion Criteria:

1. Subjects who are currently taking opioids or have used opioids in the past 14 days prior to receiving the study drug
2. Have hypersensitivity history to any opioids, naltrexone, naloxone, or related compounds or any contraindications as detailed in the OTR and OXYCONTIN tablet Summary of Product Characteristics
3. Histories of or any current conditions that might interfere with drug absorption, distribution, metabolism, or excretion
4. Subjects who are likely to have paralytic ileus or acute abdomen or to require an operation on abdominal regions
5. Subjects with biliary tract diseases, pancreatitis, prostatic hypertrophy, or corticoadrenal insufficiency
6. Subjects with respiratory depression, corpulmonale, or chronic bronchial asthma
7. Any history of seizures or symptomatic head trauma
8. Subjects with abnormal liver function (values exceeding the upper limit of normal (ULN) for alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin during the Screening Phase) or abnormal renal function (values exceeding the ULN for serum creatinine during the Screening Phase). Note: if the values of ALT, AST or total bilirubin are between 1 to 1.2 times of ULN and confirmed not clinically significant by the Investigators, the subject may be recruited after getting the approval from Sponsor.
9. Any other significant illness other than the primary disease of chronic pain during the 4 weeks preceding the entry into this study
10. Subjects who are unable to stop taking monoamine oxidase inhibitors during this trial period or time lapses less than 2 weeks since drug withdrawal prior to the study drug administration
11. Subjects who are currently taking tricyclic antidepressants or have used tricyclic antidepressants within 4 weeks prior to the study drug administration
12. Subjects who have used any medicinal product which inhibits Cytochrome P450 3A4 (CYP3A4) (e.g. troleandomycin, ketoconazole, gestodene, etc.) or induces CYP3A4 (e.g. glucocorticoids, barbiturates, rifampicin, etc.) within 4 weeks prior to the study drug administration
13. Subjects who have used any medicinal product which inhibits Cytochrome P450 2D6 (CYP2D6) (e.g. fluoxetine, quinidine, ritonavir, etc.) or induces CYP2D6 (e.g. dexamethasone, rifampicin, glutethimide, etc.) within 4 weeks prior to the study drug administration
14. Histories of smoking (being a smoker or an occasional smoker) within 45 days prior to the study drug administration and refusal to abstain from smoking during the study. According to World Health Organization (WHO), a smoker is defined as having smoked at least 1 cigarette per day continuously for more than 6 months and an occasional smoker is defined as having smoked for more than 4 times per week and less than 1 cigarette per day continuously for more than 6 months.
15. Subjects with histories of alcoholism or drug abuse. Alcoholism is defined as regular alcohol consumption exceeding 14 drinks/week (1 drink = 150 mL of wine or 360 mL of beer or 45 mL of hard liquor)
16. Consumption of alcoholic beverages within 48 hours before study drug administration, and refusal to abstain from alcohol for at least 48 hours after study drug administration
17. Refusal to abstain from food for 10 hours preceding and 4 hours following administration of the study drug and to abstain from caffeine or xanthine entirely during each confinement
18. Positive Hepatitis B Surface Antigen (HBsAg), anti-Hepatitis C Virus (HCV), anti-Human Immunodeficiency Virus (HIV), or syphilis antibody test result
19. Urine screening before study is positive for opioids, barbiturates, amphetamines, cocaine metabolites, methadone, benzodiazepines, phencyclidine, methamphetamine, or cannabinoids. Or alcohol breath test is positive
20. Any history of frequent nausea or emesis regardless of aetiology
21. Blood or blood products donated within 30 days prior to administration of the study drugs or anytime during the study, except as required by this protocol
22. Subjects who participated in a clinical research study within 30 days of study entry

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2017-10-15 (Actual); Study Completion 2018-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ZHU LUO, PhD, Principal Investigator — West Hospital, Sichuan University
Locations (1):
- West Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
Not this kind of plan with the study

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 38, from Jun2017 to Oct2017, from patient database, medical clinic, advertisement recruitment and etc.
Groups:
- OTR 40 Mg-OXYCONTIN 40 mg: the treatment sequence is OTR 40 mg dose first and then OXYCONTIN 40 mg dose in fasted state
- OXYCONTIN 40 Mg-OTR 40 mg: the treatment sequence is OXYCONTIN 40 mg dose first and then OTR 40 mg dose in fasted state
Period: Period 1
Arm/Group | OTR 40 Mg-OXYCONTIN 40 mg | OXYCONTIN 40 Mg-OTR 40 mg
Started | 19 | 19
Completed | 18 | 19
Not Completed | 1 | 0
Period: Period 2
Arm/Group | OTR 40 Mg-OXYCONTIN 40 mg | OXYCONTIN 40 Mg-OTR 40 mg
Started | 18 | 19
Completed | 16 | 17
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- OTR 40 Mg-OXYCONTIN 40 mg: the treatment sequence is OTR 40 mg dose first and then OXYCONTIN 40 mg dose
- OXYCONTIN 40 Mg-OTR 40 mg: the treatment sequence is OXYCONTIN 40 mg dose first and then OTR 40 mg dose
- Total: Total of all reporting groups
Arm/Group | OTR 40 Mg-OXYCONTIN 40 mg | OXYCONTIN 40 Mg-OTR 40 mg | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (9.61) | 40.2 (10.18) | 40.8 (9.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 8 | 5 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  HAN | 19 | 19 | 38
Weight [Mean (Standard Deviation); unit: kg] — Population: 1 subject early discontinued pre-dose because of AE
  kg
    number analyzed (Participants) | 19 | 18 | 37
    (all) | 57.87 (7.182) | 55.19 (8.088) | 56.57 (7.650)
Height [Mean (Standard Deviation); unit: cm] — Population: 1 subject early discontinued pre-dose because of AE
  cm
    number analyzed (Participants) | 19 | 18 | 37
    (all) | 160.4 (9.10) | 157.7 (8.21) | 159.1 (8.67)
BMI [Mean (Standard Deviation); unit: kg/m2] — Population: 1 subject early discontinued pre-dose because of AE
  kg/m2
    number analyzed (Participants) | 19 | 18 | 37
    (all) | 22.52 (2.419) | 22.16 (2.433) | 22.34 (2.399)

OUTCOME MEASURES:

1. Primary Outcome: Cmax of OTR Tablet 40 mg and OXYCONTIN Tablet 40 mg in a Fasted State
Description: The analysis was for PK parameters Cmax of analyte oxycodone. Analysis of Variance (ANOVA) with fixed effect terms for treatment, period, sequence, and subject within sequence for ratio of means (using log scale) were used to compare the test and the reference treatments.
Time Frame: up to 32 hours
Measure: Mean (90% Confidence Interval); unit: ng/mL
Groups:
- Cmax of OTR 40 mg: OTR Tablet 40 mg
- Cmax of OXYCONTIN® 40 mg: OXYCONTIN® Tablet 40 mg
Arm/Group | Cmax of OTR 40 mg | Cmax of OXYCONTIN® 40 mg
Number analyzed (Participants) | 32 | 32
ng/mL | 60.98 [48.336 to 73.624] | 52.23 [43.284 to 61.176]

2. Primary Outcome: AUCt of OTR Tablet 40 mg and OXYCONTIN Tablet 40 mg in a Fasted State
Description: The analysis was for PK parameters AUCt of analyte oxycodone. Analysis of Variance (ANOVA) with fixed effect terms for treatment, period, sequence, and subject within sequence for ratio of means (using log scale) were used to compare the test and the reference treatments.
Time Frame: up to 32 hours
Measure: Mean (90% Confidence Interval); unit: ng*h/ml
Groups:
- AUCt of OTR Tablet 40 mg: OTR Tablet 40 mg
- AUCt of OXYCONTIN Tablet 40 mg: OXYCONTIN Tablet 40 mg
Arm/Group | AUCt of OTR Tablet 40 mg | AUCt of OXYCONTIN Tablet 40 mg
Number analyzed (Participants) | 32 | 32
ng*h/ml | 604.5095 [485.26446 to 723.75454] | 588.6874 [478.67315 to 698.70165]

3. Primary Outcome: AUCINF of OTR Tablet 40 mg and OXYCONTIN Tablet 40 mg in a Fasted State
Description: The analysis was for PK parameters AUCINF for analyte oxycodone. Analysis of Variance (ANOVA) with fixed effect terms for treatment, period, sequence, and subject within sequence for ratio of means (using log scale) was used to compare the test and the reference treatments.
Time Frame: up to 32 hours
Measure: Mean (90% Confidence Interval); unit: ng*h/ml
Groups:
- AUCINF of OTR Tablet 40 mg: OTR Tablet 40 mg
- AUCINF of OXYCONTIN Tablet 40 mg: OXYCONTIN Tablet 40 mg
Arm/Group | AUCINF of OTR Tablet 40 mg | AUCINF of OXYCONTIN Tablet 40 mg
Number analyzed (Participants) | 32 | 32
ng*h/ml | 610.9314 [488.04292 to 733.81988] | 612.8057 [490.61681 to 734.99459]

4. Secondary Outcome: Adverse Event of OTR Tablet 40 mg and OXYCONTIN Tablet 40 mg, When Given to Chinese Subjects With Chronic Pain in a Fasted State
Description: An overall summary of adverse events will be provided by treatment groups. The number and percentage of subjects reporting adverse events will be summarised by the preferred term nested within the System Organ Classification. In addition the number of reported adverse events will be summarised.
Time Frame: up to 35 days
Measure: Number; unit: TEAEs
Groups:
- Oxycodone Tamper Resistant (OTR): Oxycodone Tamper Resistant (OTR) Tablet 40 mg
  Oxycodone Tamper Resistant: Orally taking Oxycodone Tamper Resistant 40mg in fast state
Arm/Group | Oxycodone Tamper Resistant (OTR) | OXYCONTIN®
Number analyzed (Participants) | 35 | 35
TEAEs
  Number of AEs (#) | 23 | 22
  Number of TEAEs (#) | 23 | 22
  Number of relateda TEAEs | 15 | 16

5. Secondary Outcome: Number of Lab Tests With Clinical Significance
Description: Clinical laboratory data to be summarised includes haematology, blood chemistry, and urinalysis.Each parameter will be assigned an LNH classification according to whether the value is lower than (L), within (N) or higher than (H) the reference range for that parameter. Results will be summarised using shift tables to evaluate categorical changes from baseline to end of study with respect to reference range values (lower than, within, and higher than).
Time Frame: up to 35 days
Measure: Number; unit: Lab tests with clinical significance
Groups:
- Clinical Laboratory Data of OTR Tablet 40 mg: OTR Tablet 40 mg
- Clinical Laboratory Data of OXYCONTIN Tablet 40 mg: OXYCONTIN Tablet 40 mg
Arm/Group | Clinical Laboratory Data of OTR Tablet 40 mg | Clinical Laboratory Data of OXYCONTIN Tablet 40 mg
Number analyzed (Participants) | 35 | 35
Lab tests with clinical significance | 3 | 3

6. Secondary Outcome: Number of AEs Related to Vital Sign
Description: Vital sign parameters to be summarised include systolic blood pressure, diastolic blood pressure, pulse rate, respiration rate, and axillary temperature. Vital sign results for each parameter will be assigned an LNH classification according to whether the value is lower than (L), within (N), or higher than (H) the reference range for that parameter. Vital sign results will be summarised using shift tables to evaluate categorical changes from baseline to end of study with respect to reference range values (lower than, within, and higher than).
Time Frame: up to 35 days
Measure: Number; unit: AEs of vital signs related
Groups:
- Vital Sign of OTR Tablet 40 mg: OTR tablet 40 mg
- Vital Sign of OXYCONTIN Tablet 40 mg: OXYCONTIN tablet 40 mg
Arm/Group | Vital Sign of OTR Tablet 40 mg | Vital Sign of OXYCONTIN Tablet 40 mg
Number analyzed (Participants) | 35 | 35
AEs of vital signs related | 2 | 4

7. Secondary Outcome: Number of AEs Related to ECGs
Description: Twelve-lead ECG was conducted at screening and on Day 4 of Period 2.
Time Frame: up to 35 days
Measure: Number; unit: AEs of ECG related
Groups:
- ECG of OTR Tablet 40 mg: OTR Tablet 40 mg
- ECG of OXYCONTIN Tablet 40 mg: OXYCONTIN Tablet 40 mg
Arm/Group | ECG of OTR Tablet 40 mg | ECG of OXYCONTIN Tablet 40 mg
Number analyzed (Participants) | 35 | 35
AEs of ECG related | 0 | 0

8. Secondary Outcome: Number of AEs Related to Physical Examination
Description: Physical examination was conducted at screening, and on Day -1, Day 4 in each Period.
Time Frame: up to 35 days
Measure: Number; unit: AEs related to Physical examination
Groups:
- Physical Examination of OTR Tablet 40 mg: OTR Tablet 40 mg
- Physical Examination of OXYCONTIN Tablet: OXYCONTIN Tablet 40 mg
Arm/Group | Physical Examination of OTR Tablet 40 mg | Physical Examination of OXYCONTIN Tablet
Number analyzed (Participants) | 35 | 35
AEs related to Physical examination | 0 | 0

ADVERSE EVENTS:
Time Frame: Events will be recorded from the point at which the ICF is signed until 7±1 days after last oxycodone dose in the case of completion/discontinuation from the study. This includes new AEs that are reported within 7±1 days after last oxycodone dosing after the subject's completion/discontinuation visit.
Description: same with clinicaltrials.gov Definitions.
Groups:
- OTR 40 mg: Oxycodone Tamper Resistant (OTR) Tablet 40 mg
  Oxycodone Tamper Resistant: Orally taking Oxycodone Tamper Resistant 40mg in fast state
- OXYCONTIN® 40 mg: OXYCONTIN® Tablet 40 mg
  OXYCONTIN®: Orally taking OXYCONTIN® 40mg in fast state
Arm/Group | OTR 40 mg | OXYCONTIN® 40 mg
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 4/35 | 3/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTR 40 mg (N=35) | OXYCONTIN® 40 mg (N=35)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3)
Diastolic blood pressure decreased (Cardiac disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-05-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT03398278/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/78/NCT03398278/SAP_001.pdf